CLINICAL TRIAL: NCT01655368
Title: Group Intervention for Improving Stigma Coping and Empowerment of People With Mental Illness (STEM)
Acronym: STEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfgang Gaebel, Professor (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Wolfgang Gaebel, Professor, Professor Dr., Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEM
Record Dates: First submitted 2012-06-14; First posted 2012-08-01 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Schizophrenia; Depression
MeSH Terms: conditions — Schizophrenia; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional: STEM modules (Experimental): 8 sessions of psychoeducation + 3 sessions + 1 booster session of STEM module (for schizophrenia or depression)
  Interventions: Behavioral: psychotherapeutic STEM modules
- Interventional Control (Other): 11 sessions + 1 booster session of psychoeducation for schizophrenia or depression)
  Interventions: Behavioral: Interventional control of normal psychoeducational treatment

INTERVENTIONS:
Behavioral: psychotherapeutic STEM modules — psychoeducational and psychotherapeutical group intervention. 8 sessions of psychoeducation + 3 sessions + 1 booster session of STEM module for schizophrenia or depression)
  Arms: Interventional: STEM modules
Behavioral: Interventional control of normal psychoeducational treatment — 11 sessions + 1 booster session of psychoeducation (for schizophrenia or depression)
  Arms: Interventional Control

SUMMARY:
This multi-center, 2-arm interventional study within different mental health care settings (psychiatry: in-patient, day-unit and out-patient, as well as psychiatric rehabilitation) evaluates a psychotherapeutic group intervention to improve stigma coping and empowerment using a psychotherapeutic module embedded in a psychoeducational group therapy.

DETAILED DESCRIPTION:
People with mental illness suffer both from the burden of disease itself and from the social stigma related to mental illness, hence impeding their treatment (Sartorius et al. 2005, Link et al. 1999). Negative attitudes towards and discriminating behavior against people with mental illness negatively affect health care utilization, the course of disease, compliance, self-esteem, and social functioning (Sirey et al. 2001, Link et al. 2001, Perlick et al. 2001). Internalizing negative social stereotypes (self-stigmatization; Ritsher et al. 2003, Watson et al. 2007) impairs the quality of life and leads to social withdrawal (Rüesch 2005). Furthermore, self stigma is associated with lower empowerment (Ritsher et al. 2004), a poorer social network (Lysaker et al. 2007), lower compliance (Fung et al. 2008) and a higher extent of symptoms (Corrigan et al. 2006). The stigma of mental illness leads to an impaired pursuance of individual life goals, as job-related ambitions or living in a relationship (Rüesch 2005).

Current approaches targeting the stigma of mental illness primarily focus on education about mental illness in different target groups (e.g. Gaebel et al. 2003, 2004) and can be successful, if appropriately implemented (Gaebel et al. 2008). Yet there is a lack of RCT-tested psychotherapeutic approaches which directly address patients with mental illness improving their skills of coping with stigma and discrimination. Therefore it is intended to develop, manualise, and to evaluate such a psychotherapeutic group intervention within a randomized clinical control group design.

In this context, group-based cognitive-behavioral psychotherapy has been proved as efficient therapeutic approach for patients with depression (cf. McDermut et al. 2006) and with schizophrenia (cf. Lawrence et al. 2006, Barrowclough et al. 2006) in different settings. Patients can serve each other as role models and will modify negative self-related cognitions, thus developing new cognitions supporting self-esteem (Corrigan et al. 2001). The following interventional effects should improve the patients' quality of life and also result in a reduction of frequency and length of inpatient stays and sickness-related absenteeism:

* improved skills to cope with negative stigmatizing experiences,
* a reduced burden through of self-stigmatizing cognitions,
* a better utilization of resources for disease managing in coherence with reduced self-stigmatization, and
* an improved coping with stigma-related conflicts at work.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* ICD-10 diagnosis of F2, F31.3-31.5, F32-34, F34.2, F43.2
* patients who would participate in a psychoeducational group therapy in their regular treatment
* written informed consent of the patient willing to participate
* capacity of giving consent (as diagnosed by the investigator)

Exclusion Criteria:

* insufficient knowledge of german language (reading, understanding and speaking not sufficient, as judged by the investigator)
* acute psychotic or dissociative condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
subjective quality of life | 12 months after intervention
  subjective quality of life 12 months after intervention determined by WHOQOL-BREF total score.
  To impart coping-strategies in handling stigmatization and to develop empowerment by embedding a psychotherapeutic module in psychoeducational groups.

SECONDARY OUTCOMES:
self-stigma (ISMI) | after 6 weeks, 6 months, 12 months
empowerment (BUES) | after 6 weeks, 6 months, 12 months
health care utilization (CSSRI, EQ5-D, SF-36) | after 6 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Gaebel, Prof. Dr., Principal Investigator — LVR-Klinikum Düsseldorf Kliniken der Heinrich-Heine-Universität Düsseldorf
Locations (20):
- Germany (20):
  - Klinik für Psychiatrie und Psychotherapie der RWTH, Aachen
  - Facharztpraxis Dr. Mönter, Berlin
  - Facharztpraxis Gereke, Berlin
  - Facharztpraxis Alicia Navarro Urena, Berlin
  - MediClin Bliestal Kliniken, Fachklinik für psychosomatische Medizin, Blieskastel
  - Mittelrhein-Klinik Bad Salzig der DRV, Boppard-Bad Salzig
  - Klinik für Psychiatrie und Psychotherapie, Universität zu Köln, Cologne
  - Facharztpraxis, Dr. Frosch, Düsseldorf
  - Facharztpraxis Dr. Kuhlbusch, Düsseldorf
  - LVR-Klinikum Düsseldorf - Kliniken der Heinrich-Heine Universität, Düsseldorf
  - Klinik für Psychiatrie und Psychotherapie, Uniklinik Göttingen, Göttingen
  - Klinik für Psychiatrie und Psychotherapie, UKE, Hamburg
  - Oberhavel Kliniken Hennigsdorf, Hennigsdorf
  - Berolina Klinik, Löhne
  - Klinik für Psychiatrie und Psychotherapie der Uniklinik Marburg, Marburg
  - Klinik für Psychiatrie und Psychotherapie, LMU, Munich
  - Reha-Zentrum Seehof der DRV, Teltow
  - Psychiatrisch-psychotherapeutisches Rehabilitationszentrum grund.stein, Tübingen
  - Klinik für Psychiatrie und Psychotherapie, Tübingen
  - AHG Klinik Waren, Waren

REFERENCES:
- [Background] Barrowclough C, Haddock G, Lobban F, Jones S, Siddle R, Roberts C, Gregg L. Group cognitive-behavioural therapy for schizophrenia. Randomised controlled trial. Br J Psychiatry. 2006 Dec;189:527-32. doi: 10.1192/bjp.bp.106.021386. PMID 17139037
- [Background] Corrigan P, Lundin R. Don´t call me nuts: Coping with the stigma of mental illness. Recovery Press, Chicago 2001
- [Background] Corrigan PW, Watson AC, Barr L (2006) The Self-Stigma of Mental Illness: Implications for Self-Esteem and Self-Efficacy. J Soc Clin Psychol 25: 875-884
- [Background] Gaebel W, Baumann AE. Interventions to reduce the stigma associated with severe mental illness: experiences from the open the doors program in Germany. Can J Psychiatry. 2003 Nov;48(10):657-62. doi: 10.1177/070674370304801003. PMID 14674047
- [Background] Gaebel W, Zäske H, Baumann A (2004) Stigma erschwert Behandlung und Integration. Dtsch Ärztebl 101: A3253-3255
- [Background] Gaebel W, Zaske H, Baumann AE, Klosterkotter J, Maier W, Decker P, Moller HJ. Evaluation of the German WPA "program against stigma and discrimination because of schizophrenia--Open the Doors": results from representative telephone surveys before and after three years of antistigma interventions. Schizophr Res. 2008 Jan;98(1-3):184-93. doi: 10.1016/j.schres.2007.09.013. Epub 2007 Oct 24. PMID 17961985
- [Background] Lawrence R, Bradshaw T, Mairs H. Group cognitive behavioural therapy for schizophrenia: a systematic review of the literature. J Psychiatr Ment Health Nurs. 2006 Dec;13(6):673-81. doi: 10.1111/j.1365-2850.2006.01014.x. PMID 17087669
- [Background] Link BG, Phelan JC. Labeling and stigma. In: The Handbook of the Sociology of Mental Health, Hrsg. CS Aneshensel, JC Phelan. Plenum, New York 1999
- [Background] Link BG, Struening EL, Neese-Todd S, Asmussen S, Phelan JC. Stigma as a barrier to recovery: The consequences of stigma for the self-esteem of people with mental illnesses. Psychiatr Serv. 2001 Dec;52(12):1621-6. doi: 10.1176/appi.ps.52.12.1621. PMID 11726753
- [Background] Lysaker PH, Roe D, Yanos PT. Toward understanding the insight paradox: internalized stigma moderates the association between insight and social functioning, hope, and self-esteem among people with schizophrenia spectrum disorders. Schizophr Bull. 2007 Jan;33(1):192-9. doi: 10.1093/schbul/sbl016. Epub 2006 Aug 7. PMID 16894025
- [Background] McDermut W, Miller IW, Brown RA (2006) The Efficacy of Group Psychotherapy for Depression: A Meta-analysis and Review of the Empirical Research. Clinical Psychol: Science and Practice 8: 98-116
- [Background] Perlick DA, Rosenheck RA, Clarkin JF, Sirey JA, Salahi J, Struening EL, Link BG. Stigma as a barrier to recovery: Adverse effects of perceived stigma on social adaptation of persons diagnosed with bipolar affective disorder. Psychiatr Serv. 2001 Dec;52(12):1627-32. doi: 10.1176/appi.ps.52.12.1627. PMID 11726754
- [Background] Ritsher JB, Otilingam PG, Grajales M. Internalized stigma of mental illness: psychometric properties of a new measure. Psychiatry Res. 2003 Nov 1;121(1):31-49. doi: 10.1016/j.psychres.2003.08.008. PMID 14572622
- [Background] Ritsher JB, Phelan JC. Internalized stigma predicts erosion of morale among psychiatric outpatients. Psychiatry Res. 2004 Dec 30;129(3):257-65. doi: 10.1016/j.psychres.2004.08.003. PMID 15661319
- [Background] Rusch N, Corrigan PW, Wassel A, Michaels P, Larson JE, Olschewski M, Wilkniss S, Batia K. Self-stigma, group identification, perceived legitimacy of discrimination and mental health service use. Br J Psychiatry. 2009 Dec;195(6):551-2. doi: 10.1192/bjp.bp.109.067157. PMID 19949209
- [Background] Rüesch P. Soziale Netzwerke und Lebensqualität. In: Gaebel W, Möller HJ, Rössler W (Hrsg). Stigma - Diskriminierung - Bewältigung. Kohlhammer, Stuttgart 2005
- [Background] Sartorius N, Schulze H. Reducing the stigma of mental illness. Cambridge University Press, Cambridge 2005
- [Background] Sirey JA, Bruce ML, Alexopoulos GS, Perlick DA, Friedman SJ, Meyers BS. Stigma as a barrier to recovery: Perceived stigma and patient-rated severity of illness as predictors of antidepressant drug adherence. Psychiatr Serv. 2001 Dec;52(12):1615-20. doi: 10.1176/appi.ps.52.12.1615. PMID 11726752
- [Background] Watson AC, Corrigan P, Larson JE, Sells M. Self-stigma in people with mental illness. Schizophr Bull. 2007 Nov;33(6):1312-8. doi: 10.1093/schbul/sbl076. Epub 2007 Jan 25. PMID 17255118
- [Derived] Gaebel W, Zaske H, Hesse K, Klingberg S, Ohmann C, Grebe J, Kolbe H, Icks A, Schneider F, Backes V, Wolff-Menzler C, Guse B, Gallinat J, Bock T, Jockers-Scherubl MC, Kruger T, Jessen F, Bechdolf A, Kircher T, Konrad C, Falkai P, Schaub A, Rudolph M, Kollner V, Schmid-Ott G, Linden M, Lieberei B, Stuhlinger M, Sommerfeld S, Schumacher A, Krenge S, Gereke S, Monter N, Navarro-Urena A, Frosch G, Kuhlbusch FJ, Cleveland H, Riesbeck M. Promoting stigma coping and empowerment in patients with schizophrenia and depression: results of a cluster-RCT. Eur Arch Psychiatry Clin Neurosci. 2020 Aug;270(5):501-511. doi: 10.1007/s00406-019-01064-3. Epub 2019 Sep 13. PMID 31520149
- See also: homepage of the responsible party — http://www.rk-duesseldorf.lvr.de